CLINICAL TRIAL: NCT01723332
Title: The CHAPTER II Study - Congenital Heart Adolescents Participating in Transition Evaluation Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Andrew Mackie, Associate Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHAPTER II
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Congenital Heart Disease
Keywords: Transition from pediatric to adult clinical care
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Clinical based educational and self management intervention.
  Interventions: Behavioral: Educational; Behavioral: Self management
- Usual Care (No Intervention): Youth seen in the Cardiology clinic see a nurse only to measure weight, height, and blood pressure. They rely on their cardiologist for information about their heart condition. The approach and amount of time taken by each cardiologist with a youth varies.

INTERVENTIONS:
Behavioral: Educational — The first interaction will happen at study enrolment and will be educational in nature.
  Following the session, the nurse will follow up with the participant to discuss any questions.
  Arms: Intervention
Behavioral: Self management — The second interaction will take place 2 months after enrollment and will focus on self management and communication skills.
  Following the session, the nurse will follow up with the participant to discuss any questions.
  Arms: Intervention

SUMMARY:
Transition is the planned movement of teens with chronic conditions from child-centered to adult-oriented healthcare. National bodies have published detailed guidelines about the importance of helping teens move to adult healthcare. However, there is no research regarding how to best organize and deliver Congenital Heart Disease (CHD) transition programs. Data is urgently needed. Therefore, the aim of this program is to develop research evidence that will better prepare health care providers to improve how they can help adolescents with transition.

This project will determine whether a nurse-led transition intervention program is better at preparing teens with CHD to independently manage their medical care, compared to the care that is currently provided. The most important finding of this study will be whether or not these teens subsequently attend the adult cardiology clinic that specializes in CHD problems, and the timing of when they attend.

Hypothesis: A transition intervention in combination with usual care, improved time to first Adult Congenital Heart Disease (ACHD) clinic attendance compared to usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* 16 and 17 year olds with moderate or complex CHD

Exclusion Criteria:

* Significant developmental delay
* Previous heart transplantation

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2012-11; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Excess time to first ACHD clinic appointment. | 12 - 24 months post enrolment

SECONDARY OUTCOMES:
Change in adolescent knowledge of their condition. | 6 - 18 months post enrolment
Change in adolescent's self-management and self-advocacy skills/ | 6 - 18 months post enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Mackie, MD, SM, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Hospital For Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Mackie AS, Rempel GR, Kovacs AH, Kaufman M, Rankin KN, Jelen A, Yaskina M, Sananes R, Oechslin E, Dragieva D, Mustafa S, Williams E, Schuh M, Manlhiot C, Anthony SJ, Magill-Evans J, Nicholas D, McCrindle BW. Transition Intervention for Adolescents With Congenital Heart Disease. J Am Coll Cardiol. 2018 Apr 24;71(16):1768-1777. doi: 10.1016/j.jacc.2018.02.043. PMID 29673467
- [Derived] Mackie AS, Rempel GR, Kovacs AH, Kaufman M, Rankin KN, Jelen A, Manlhiot C, Anthony SJ, Magill-Evans J, Nicholas D, Sananes R, Oechslin E, Dragieva D, Mustafa S, Williams E, Schuh M, McCrindle BW. A cluster randomized trial of a transition intervention for adolescents with congenital heart disease: rationale and design of the CHAPTER 2 study. BMC Cardiovasc Disord. 2016 Jun 6;16:127. doi: 10.1186/s12872-016-0307-2. PMID 27266868